CLINICAL TRIAL: NCT05125718
Title: Clinical and Metagenomic Investigation of Locally Delivered Synthetic Antimicrobial Peptide Gel in Non-surgical Periodontal Treatment: a Pilot Study.
Brief Title: Clinical and Metagenomic Investigation of Antimicrobial Peptide Gel in Periodontal Treatment.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Tan Hooi Shan, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMP-01
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: split-mouth study
Who Masked: Participant, Care Provider
Masking Description: blinding of subject and clinician
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (antimicrobial peptide) (Experimental): Half of the dentition will receive scaling and root surface debridement within a week followed by the application of antimicrobial peptide gel Ace Helper™ into the site with pocket depth >5mm until overflow noticed. Antimicrobial peptide (AMP) will be reapplied for 2 more times at an interval of 3 days. Antimicrobial peptide gel Ace Helper™ contained 0.85% synthetic AMP (TAPS-18) designed based on the basic structure of cathelicidin, hydroxyethyl cellulose, and purified water.
  Interventions: Drug: 0.85% synthetic antimicrobial peptide TAPS-18
- control group (normal saline) (Sham Comparator): Half of the dentition will receive scaling and root surface debridement within a week followed by the irrigation of 0.9% normal saline into the site with pocket depth >5mm. Normal saline irrigation will be repeated for 2 more times at an interval of 3 days.
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: 0.85% synthetic antimicrobial peptide TAPS-18 — commercially available synthetic antimicrobial peptide gel for periodontal disease treatment
  Other Names: antimicrobial peptide gel Ace Helper™
  Arms: test group (antimicrobial peptide)
Drug: 0.9% normal saline — commercially available normal saline Sodium Chloride irrigation solution
  Other Names: RinsCap Normal Saline Sodium Chloride Irrigation Solution
  Arms: control group (normal saline)

SUMMARY:
Background and objective(s): Periodontitis is initiated by a dysbiotic host-microbe relationship. Standard periodontal treatment involves oral hygiene education, mechanical debridement and periodic follow-ups with the aims of pocket closure and maintaining a symbiotic microbial community. Nonetheless, this therapy alone may fail due to the limitations of mechanical instrumentation. The use of antimicrobial in combination to subgingival debridement has been proposed for initial and recurrent periodontitis to enhance the effectiveness of mechanical instrumentation. Antimicrobial peptide (AMP) comprised of a wide range of peptide, was found naturally in various life forms or manufactured as a synthetic compound. This study was conducted to evaluate the use of AMP as an adjunct to non-surgical periodontal treatment in terms of clinical and microbiological outcomes.

Hypothesis

• There are changes in clinical periodontal parameters and subgingival microbial profile following treatment with locally delivered synthetic AMP.

DETAILED DESCRIPTION:
study design: This was a split-mouth randomised pilot study of a 3-months follow-up.

Sample size calculation: The sample size was calculated using G*Power software version 3.1.9.4 (Franz Faul, Universitat Kiel, Germany). Estimation of sample size was based on the mean and standard deviation of CAL between the test and control group of previous publication (Singh et al., 2018). Four samples in each group (test and control) were required to achieve 80% power at a significant level of 5%.

Randomisation: The random allocation sequence was generated by another person who was not directly involved in the study using a Research Randomizer tools (https://www.randomizer.org/). Periodontal sites of each patient were randomised at a split mouth level (left or right halves of the dentition) to one of the two treatment groups. Allocated treatments were inserted into an opaque envelop. Treatment allocation was concealed from the clinician and only revealed once subgingival debridement was completed.

intervention: At baseline, clinical measurement was recorded and target sites (sites with PPD ≥6mm) were identified. subgingival plaque were collected at target sites. The same clinician performed full mouth scaling and subgingival debridement, coupled with standardised oral hygiene instruction for all subjects. Upon the completion of treatment, second clinician applied the treatments according to the randomisation.

* Test group: Subgingival instrumentation followed by Antimcrobial peptide gel (AMP) application in all target sites.
* Control group: Subgingival instrumentation and normal saline irrigation in all target sites.

Test and control intervention will be repeated for another 2 applications at an interval of 3 days. Subjects were re-examined and plaque sampling will be repeated at 6 weeks and 12 weeks.

statistical analysis: Clinical parameters were reported as mean and standard deviation. P-value <0.05 was considered statistically significant. intergroup and intragroup comparison of mean bleeding score, pocket depth, clinical attachment level will be conducted using SPSS software. For the metagenomic data, alpha and beta diversity were computed using QIIME 2. The difference in the relative abundance of individual genus over time will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* • Subject diagnosed with generalised periodontitis Stage III of any grade (Caton et al., 2018).

  * Age ≥21 years old.
  * Subject is in good general health without any remarkable past history of disease except for well controlled diabetes (HbA1c ≤6.5%) (Clinical practice guidelines on management of type 2 diabetes mellitus., 2020).
  * Presence of at least 20 teeth.
  * Presence of at least 2 non-adjacent sites located in contralateral quadrant with interproximal probing pocket depth (PPD) ≥6mm.

Exclusion Criteria:

* • Received subgingival scaling in the previous 6 months.

  * Use of antibiotic in the past 6 months.
  * Taking steroidal and non-steroidal anti-inflammatory agents on a daily basis.
  * Medical condition requiring antibiotic prophylaxis.
  * Pregnancy or lactating.
  * Smoking ≥10 cigarettes per day.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
clinical measurement of pocket depth (mm) | 6 weeks and 12 weeks
  changes in pocket depth after the test and control intervention. pocket depth is measured from the gingival margin to base of pocket using UNC-15 probe
clinical measurement of clinical attachment level (mm) | 6 weeks and 12 weeks
  changes in clinical attachment level after the test and control intervention. clinical attachment level is measured from cemento-enamel junction to base of pocket using UNC-15 probe.
metagenomic analysis of the relative abundance (%) of bacterial from subgingival plaque | 6 weeks and 12 weeks
  changes in relative abundance of bacterial after the test and control intervention is measured by the metagenomic analysis using subgingival plaque

CONTACTS AND LOCATIONS:
Overall Officials: Hooi Shan, Principal Investigator — faculty of dentistry, University of Malaya
Locations (1):
- faculty of dentistry, University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No